CLINICAL TRIAL: NCT01710332
Title: Intravitreal Aflibercept Injection for Persistent Central Serous Chorioretinopathy: A Prospective Pilot Study
Brief Title: The Safety & Efficacy of Intravitreal Aflibercept Injection in Patients With Persistent Central Serous Chorioretinopathy
Acronym: CONTAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Allen C. Ho, MD, Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSRII; 20121564 (Other: Western IRB)
Record Dates: First submitted 2012-10-16; First posted 2012-10-19 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-05

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Persistent; Central; Serous; Chorioretinopathy; Regeneron; CSR; CSCR
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravitreal Aflibercept Injection (x4) (Experimental): 2 mg / Intravitreal / every 1 month x 3 months and at month 4 (Drug administered 4 times).
  Interventions: Drug: Intravitreal Aflibercept Injection
- Intravitreal Aflibercept Injection (x6) (Experimental): 2 mg / Intravitreal / every 1 month x 6 months ((Drug administered 6 times).
  Interventions: Drug: Intravitreal Aflibercept Injection

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection — GROUP A - Aflibercept 2 mg injected at Baseline, Month 1, Month 2, and Month 4 (four injections total).
  GROUP B - Aflibercept 2 mg injected at Baseline, Month 1, Month 2, Month 3, Month 4, and Month 5 (six injections total).
  Other Names: Eylea

SUMMARY:
A preliminary study to determine the safety and efficacy of intravitreal aflibercept injection in patients with persistent central serous chorioretinopathy.

DETAILED DESCRIPTION:
Intravitreal Aflibercept Injection for Persistent Central Serous Chorioretinopathy: A Prospective Pilot Study

ELIGIBILITY:
Inclusion Criteria:

* Pre-treatment acuity of 20/40- 20/320
* Macular fluid on optical coherence tomography for greater than 3 months
* Leakage on fluorescein angiography
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent

Exclusion Criteria:

* Treatment for CSCR in the study eye (anti-VEGF, PDT, or laser) within three months prior to study enrollment
* Presence of choroidal neovascularization on enrollment imaging
* Prior vitrectomy in the study eye
* Presence of any substantial ocular disease (other than CSCR) that may compromise vision in the study eye and /or confound interpretation of the data; e.g. substantial cataracts, advanced glaucoma, optic neuritis, optic neuropathy or atrophy, marked macular atrophy, ocular vascular occlusion, history of retinal detachment, uveitis, viral or other forms of chorioretinitis, etc.
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Uncontrolled glaucoma in the study eye (defined as IOP ≥ 25 mmHg despite treatment with anti-glaucoma medication)
* Active ocular infection or inflammation in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Prior treatment with systemic anti-VEGF agents
* Cerebrovascular accident or myocardial infarction within the preceding 6 months.
* History of allergy to fluorescein, povidone iodine (Betadine) or aflibercept
* Participation in a study of an investigational drug or device within 30 days prior to potential enrollment into the study
* Pregnant or breast-feeding women Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

  * Contraception is not required for men with documented vasectomy.

    * Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Ho, MD, Principal Investigator
Locations (2):
- United States (2):
  - Mid Atlantic Retina- Huntingdon Valley, Huntingdon Valley, Pennsylvania
  - Mid Atlantic Retna- Wills Eye Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203
- [Derived] Pitcher JD 3rd, Witkin AJ, DeCroos FC, Ho AC. A prospective pilot study of intravitreal aflibercept for the treatment of chronic central serous chorioretinopathy: the CONTAIN study. Br J Ophthalmol. 2015 Jun;99(6):848-52. doi: 10.1136/bjophthalmol-2014-306018. Epub 2015 Jan 16. PMID 25595177

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravitreal Aflibercept Injection (x4): 2 mg / Intravitreal / every 1 month x 3 months and at month 4 (Drug administered 4 times).
  Intravitreal Aflibercept Injection: GROUP A - Aflibercept 2 mg injected at Baseline, Month 1, Month 2, and Month 4 (four injections total).
  GROUP B - Aflibercept 2 mg injected at Baseline, Month 1, Month 2, Month 3, Month 4, and Month 5 (six injections total).
- Intravitreal Aflibercept Injection (x6): 2 mg / Intravitreal / every 1 month x 6 months ((Drug administered 6 times).
  Intravitreal Aflibercept Injection: GROUP A - Aflibercept 2 mg injected at Baseline, Month 1, Month 2, and Month 4 (four injections total).
  GROUP B - Aflibercept 2 mg injected at Baseline, Month 1, Month 2, Month 3, Month 4, and Month 5 (six injections total).
Period: Overall Study
Arm/Group | Intravitreal Aflibercept Injection (x4) | Intravitreal Aflibercept Injection (x6)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravitreal Aflibercept Injection (x4) | Intravitreal Aflibercept Injection (x6) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (12.8) | 53.5 (9.6) | 53.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety of Intravitreal Aflibercept Injection
Description: Safety will be measured by the amount, significance and details of adverse events/reactions to the study drug.
Time Frame: 6 months
Measure: Number; unit: adverse events
Groups:
- Intravitreal Aflibercept Injection (x4): 2 mg / Intravitreal / every 1 month x 3 months and at month 4 (Drug administered 4 times).
  Intravitreal Aflibercept Injection: GROUP A - Aflibercept 2 mg injected at Baseline, Month 1, Month 2, and Month 4 (four injections total).
- Intravitreal Aflibercept Injection (x6): 2 mg / Intravitreal / every 1 month x 6 months ((Drug administered 6 times).
  GROUP B - Aflibercept 2 mg injected at Baseline, Month 1, Month 2, Month 3, Month 4, and Month 5 (six injections total).
Arm/Group | Intravitreal Aflibercept Injection (x4) | Intravitreal Aflibercept Injection (x6)
Number analyzed (Participants) | 6 | 6
adverse events | 0 | 0

2. Secondary Outcome: Change in Vision Based on Letter Score
Description: • Mean change from baseline in best-corrected ETDRS (Early Treatment of Diabetic Retinopathy Study) letter score
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Intravitreal Aflibercept Injection (x4) | Intravitreal Aflibercept Injection (x6)
Number analyzed (Participants) | 6 | 6
ETDRS letters | -0.3 (12.4) | 4.7 (13.4)

ADVERSE EVENTS:
Arm/Group | Intravitreal Aflibercept Injection (x4) | Intravitreal Aflibercept Injection (x6)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No